CLINICAL TRIAL: NCT01857401
Title: Development of a Novel Human In Vitro Sarcoidosis Model
Status: Completed | Type: Observational
Sponsor: Elliott Crouser MD (Other)
Responsible Party: Sponsor-Investigator, Elliott Crouser MD, Assistant Professor of Internal Medicine, Ohio State University
Organization: Ohio State University (Other)
Other Study IDs: 2012H0073
Record Dates: First submitted 2013-05-02; First posted 2013-05-20 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-11

CONDITIONS: Sarcoidosis
MeSH Terms: conditions — Sarcoidosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational study: Blood draw only, observational study
  Interventions: Other: No intervention, observational study only

INTERVENTIONS:
Other: No intervention, observational study only — No intervention. We are collecting blood for an ex vivo study

SUMMARY:
There is currently no experimental model that accurately represents sarcoidosis. The lack of a useful research model significantly slows progress towards developing new treatments for sarcoidosis. The investigators plan to develop a new model for sarcoidosis research and will test the model to see if it helps us understand how sarcoidosis develops and if it is useful for testing new treatments.

DETAILED DESCRIPTION:
Sarcoidosis is a systemic granulomatous disease of unknown cause, most commonly affecting the lungs, which tends to afflict young adults in the prime of their lives. Recent data indicating that sarcoidosis mortality rates are rising in the U.S. (1) and Europe (2) highlight the inadequacy of current therapies. As noted in a recent NIH-sponsored sarcoidosis workshop, the lack of relevant animal, computer or in vitro models represents a bottleneck for progress towards understanding disease mechanisms and developing highly effective sarcoidosis treatments (3). The lack of useful disease models likely contributes to the current lack (zero) of investigator-initiated (RO1) projects supporting sarcoidosis research.

The long-term goal of this proposal is to develop a novel human sarcoidosis research model to fill the current void in the field, thereby expediting exploration of basic disease mechanisms and pre-clinical testing of novel therapies. The objective of this application, which is the first step towards achieving the long-term goal, is to develop a novel in vitro human granuloma model to represent abnormal granuloma formation in the context of sarcoidosis. In this regard, a growing body of evidence indicates that mycobacterial antigens are commonly harbored in sarcoidosis tissues, to which these patients are sensitized (4, 5). Our central hypothesis is that the pathological mechanisms of sarcoidosis can be modeled in vitro, as represented by abnormal granuloma formation in response to mycobacterial and other ubiquitous environmental antigens. The feasibility of our proposed model is supported by preliminary studies showing that subjects sensitized to Mycobacterium tuberculosis antigens (latent TB tuberculosis with a positive TB skin test) form well-organized granulomas readily in response to challenge with TB antigens, compared to healthy controls. This project is highly innovative and we feel has an excellent likelihood of leading to a critical breakthrough in the field of sarcoidosis research.

ELIGIBILITY:
Inclusion Criteria:

* sarcoidosis, subjects (18 - 45 years of age), including 30 sarcoidosis, 15 latent TB and 15 healthy controls.

Exclusion Criteria:

* pregnant women

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: primary care clinic
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-12-19 (Actual); Primary Completion 2017-02-02 (Actual); Study Completion 2017-02-02 (Actual)

PRIMARY OUTCOMES:
Sarcoidosis patients, volunteers with latent TB, and healthy volunteer subjects will be recruited to donate peripheral blood for isolation of peripheral blood mononuclear cells. | 2-4 years
  We hypothesize that patients with the active sarcoidosis phenotype will exhibit accelerated granuloma formation with higher IL-10(IL Interleukin)and IL-4 expression relative to patients with the self-limited sarcoidosis phenotype

CONTACTS AND LOCATIONS:
Overall Officials: Elliott Crouser, MD, Principal Investigator — Ohio State University
Locations (1):
- Biomedical Research Tower, 10th floor, Columbus, Ohio, United States

REFERENCES:
- [Derived] Locke LW, Crouser ED, White P, Julian MW, Caceres EG, Papp AC, Le VT, Sadee W, Schlesinger LS. IL-13-regulated Macrophage Polarization during Granuloma Formation in an In Vitro Human Sarcoidosis Model. Am J Respir Cell Mol Biol. 2019 Jan;60(1):84-95. doi: 10.1165/rcmb.2018-0053OC. PMID 30134122
- [Derived] Crouser ED, White P, Caceres EG, Julian MW, Papp AC, Locke LW, Sadee W, Schlesinger LS. A Novel In Vitro Human Granuloma Model of Sarcoidosis and Latent Tuberculosis Infection. Am J Respir Cell Mol Biol. 2017 Oct;57(4):487-498. doi: 10.1165/rcmb.2016-0321OC. PMID 28598206